CLINICAL TRIAL: NCT01884779
Title: Histoplasmosis in the Guiana Shield and the French West Indies: Evaluating Prevalence in HIV + Patients with a Rapid Diagnostic Test Using an ELISA Capture Method for the Detection of Histoplasma Antigens in Blood and Urine.
Brief Title: Prevalence of Histoplasmosis in HIV + Patients with a Rapid Diagnostic Test in West Indies
Acronym: EDIRAPHIS
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12260 EDIRAPHIS
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: HIV; Histoplasmosis; Histoplasma capsulatum var.capsulatum; ELISA test
MeSH Terms: conditions — Histoplasmosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Urine, serum and Histoplasma capsulatum var. capsulatum strains
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Histoplasma capsulatum var. capsulatum histoplasmosis is the leading cause of acquired immunodeficiency syndrome (AIDS) and death in French Guiana and probably in the Amazon. The diagnosis of this disease requires invasives procedures, laboratory performance, and delays up to several weeks. The Mycotic Diseases Branch of the Centers for Disease Control and Prevention (CDC) has established a rapid, sensitive and specific ELISA test for blood and urine samples that looks interesting in endemic areas, particularly in developing countries. The study aims to measure the proportion of HIV-infected patients hospitalized or in outpatient awaiting hospitalization for a suspicion of infectious syndrome whose serum and/or urinary antigen detection tests are positive for Histoplasma capsulatum var. capsulatum.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or over).
* Patient seen while hospitalized or in outpatient awaiting hospitalization.
* HIV1 or HIV2 infection confirmed by techniques validated in France and in Suriname, either before the episode considered, or discovered concomitantly.
* Patient presenting at least one of the three followings items: an alteration of their general condition (with a grade 1 according to the WHO Performance Status scale) and/or a fever and/or symptoms suggestive of an infectious syndrome.
* Medical prescription for the collection of blood and urine specimens to test for an infectious agent within 7 days following admission to the hospital.
* Written consent to participate in the study obtained.

Exclusion Criteria:

* Refusal to participate in the study.
* Patient in a critical condition that doesn't allow physicians to get an informed consent without a legal representative to represent him and sign a consent form for the patient participation in the study.
* Ongoing antifungal treatment or antifungal treatment stopped during the month preceding the inclusion date (topic antifungal therapy not considered at this point).
* Patient in detention at the time of admission to the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (aged 18 or over), seen while hospitalized or in outpatient awaiting hospitalization, HIV1 or HIV2 infection confirmed by techniques validated in France and in Suriname, either before the episode considered, or discovered concomitantly, and presenting at least one of the three followings items: an alteration of their general condition (with a grade 1 according to the WHO Performance Status scale) and/or a fever and/or symptoms suggestive of an infectious syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 727 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-11-03 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-infected patients hospitalized or in outpatient awaiting hospitalization for a suspicion of infectious syndrome whose serum and/or urinary antigen detection tests are positive for Histoplasma capsulatum var. capsulatum. | At the time of inclusion (baseline)

SECONDARY OUTCOMES:
Sensitivity of the ELISA test on urine and blood specimens | At the time of inclusion (baseline)
Sensibility of the ELISA test on urine and blood specimens | At the time of inclusion (baseline)
Negative predictive value of the ELISA test on urine and blood specimens | At the time of inclusion (baseline)
Comparison of the distribution of Histoplasma antigen concentrations in urine and serum specimens according to severity of cases of histoplasmosis due to Histoplasma capsulatum var. capsulatum | At the time of inclusion (baseline)
Comparison of the socio-demographic, clinical, paraclinical and therapeutic characteristics according to severity of cases of histoplasmosis due to Histoplasma capsulatum var. capsulatum | 30 days or 90 days after inclusion
Comparison of the factors for environmental exposure to Histoplasma capsulatum var capsulatum between patients with a positive ELISA test and/or fungal culture for histoplasmosis and those who tested negative for histoplasmosis | At the time of inclusion
Frequency of histoplasmosis compared to the other main diagnoses according to three sets of comparisons: positive ELISA test and positive fungal culture; positive ELISA test and negative fungal culture; negative ELISA test and positive fungal culture | 90 days after inclusion
Comparison of the socio-demographic, clinical, paraclinical, therapeutic and survival outcome characteristics of cases of histoplasmosis compared to those who tested negative for histoplasmosis | 90 days after inclusion
Identify the prognostic factors for short-term unfavourable progression of cases of histoplasmosis due to Histoplasma capsulatum var. capsulatum confirmed by ELISA test and/or by fungal culture | 30 days and 90 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu NACHER, MD, PhD, Study Chair — CIE 802 Inserm / DGOS; Stephen G VREDEN, MD, PhD, Study Chair — Foundation for Scientific Research Suriname (SWOS)
Locations (7):
- France (4):
  - Pointe-à-Pitre University Hospital, Pointe à Pitre, Guadeloupe
  - Cayenne General Hospital, Cayenne, Guyane
  - Western French Guiana Hospital, Saint-Laurent-du-Maroni, Guyane
  - Fort-de-France University Hospital, Fort-de-France, Martinique
- Suriname (3):
  - 's Lands Hospital, Paramaribo, Paramaribo District
  - Academisch Ziekenhuis Paramaribo Hospital, Paramaribo, Paramaribo District
  - Diakonessenhuis hospital, Paramaribo, Paramaribo District